CLINICAL TRIAL: NCT03404297
Title: Evaluation of Locally-sourced Compression Therapy for Treatment of Chronic Leg Ulcers and Management of Kaposi Sarcoma Leg Lymphedema in Western Kenya
Brief Title: Compression Therapy for Leg Ulcers and Kaposi Sarcoma in Western Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of California, San Francisco (Other); Moi Teaching and Referral Hospital (Other); Moi Univeristy (Other); Purdue University (Other); Indiana Clinical and Translational Sciences Institute (Other)
Responsible Party: Principal Investigator, Sonak Pastakia, Professor of Pharmacy, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1710769547
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Leg Ulcer; Kaposi Sarcoma; HIV/AIDS and Infections
Keywords: compression therapy; Kenya; Kaposi Sarcoma; Locally sourced; wrapping; chronic leg ulcers
MeSH Terms: conditions — Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Infections

STUDY DESIGN:
Intervention Model Description: The study will include two different types of evaluation based on the disease process that the patient has. For patients with chronic leg ulcers, a retrospective, observational approach will be used to track the efficacy of locally sourced compression in improving wound healing.
  For patients with Kaposi Sarcoma associated leg lymphedema, they will be randomized to to receive immediate compression therapy or delayed compression therapy.
Masking Description: The trial is open label but the randomization scheme will be determined by an automatic randomization algorithm performed independently of the investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Compression Therapy Arm (Experimental): Patients in this arm will receive a locally sourced version of compression therapy while concurrently receiving chemotherapy
  Interventions: Other: Locally sourced compression therapy
- Delayed Compression Therapy Arm (Placebo Comparator): Patients in this arm will receive a locally sourced version of compression therapy after completing ~ 14 weeks of chemotherapy.
  Interventions: Other: Locally sourced compression therapy

INTERVENTIONS:
Other: Locally sourced compression therapy — The dressing is made up of a zinc oxide impregnated compression wrapping

SUMMARY:
The efficacy of locally sourced compression therapy in the management of chronic leg ulcers and Kaposi Sarcoma in western Kenya will be studied in a rural setting

DETAILED DESCRIPTION:
Compression therapy is a well-established cornerstone therapy and part of routine clinical care for chronic leg ulcers from venous disease and lymphedema, including Kaposi sarcoma (KS)-associated lymphedema. Chronic leg ulcers, from trauma or chronic venous disease, and lymphedema have a significant impact on quality of life, driven by pain, foul odor, and restricted mobility. The provision of compression therapy in resource-limited settings, as in western Kenya and other regions of East Africa, is a major challenge. In western Kenya, locally available elastic stockings are priced at 10-15 USD (1000-1500 kshs) per pair. Pre-packaged brand name kits are not locally available or affordable for patients, as imported kits costs 7-20 USD (700-2000 kshs) per package. However, materials used routinely in wound care, namely elastic crepe, gauze, and zinc oxide, are readily available and affordable for patients. Supplies required to dress one affected leg for a week cost 2 USD (200 kshs). The use of locally-sourced routine wound care supplies for compression therapy is poised to have significant impact on reducing morbidity, social stigma, and economic loss associated with chronic leg ulcers and Kaposi sarcoma-associated lymphedema. Demonstration of its feasibility and efficacy in treating chronic leg ulcers and Kaposi sarcoma-associated lymphedema in western Kenya could have far-reaching implications for the treatment of these prevalent conditions across East Africa and sub-Saharan Africa. This project will utilize a 1) retrospective study design to evaluate the efficacy of compression therapy for the treatment of chronic leg ulcer patients seen at Turbo Health Center, one of the Academic Model for Providing Access to Healthcare (AMPATH) sites and 2) randomized controlled trial to evaluate the efficacy of compression therapy in the management of Kaposi sarcoma leg lymphedema patients seen at AMPATH/MTRH oncology clinics. If the outcomes of this project support the use of locally-sourced compression therapy in the treatment of chronic leg ulcers and Kaposi sarcoma-associated lymphedema, future studies for chronic leg ulcers will focus on scaling up use of locally-sourced compression therapy at other AMPATH clinics and exploring feasibility of community-based care. Future studies for Kaposi sarcoma lymphedema will focus on exploring feasibility of community or home-based lymphedema care.

ELIGIBILITY:
Retrospective Chronic Leg Ulcer Arm Investigation

Inclusion Criteria:

* Older than 18 years of age
* Received paste bandage compression therapy as part of routine wound care
* Presence of venous ulcer for more than 6 weeks. Venous ulcer defined as a wound of the lower extremity in an individual with adequate lower extremity arterial flow located in the gaiter region of the leg (between the knee and ankle) with clinical signs of venous disease (edema, varicose veins) (19) OR
* Presence of trauma-related ulcer for more than 6 weeks

Exclusion Criteria:

* Patients with peripheral arterial disease as documented via documented history or peripheral vascular physical examination. (20)
* Patients diagnosed with diabetic foot ulcers
* Patients diagnosed with ulcers from inflammatory conditions (pyoderma gangrenosum, vasculitis, rheumatoid arthritis, and other connective tissue diseases/autoimmune diseases)
* Concomitant diagnosis of decompensated heart failure, acute phase dermatitis (at the time of the study), acute phase deep vein thrombosis

Prospective Kaposi Sarcoma Investigation

Inclusion Criteria:

* Older than 18 years of age
* Diagnosis of biopsy-proven Kaposi sarcoma with associated leg lymphedema
* Leg lymphedema consistent with Campisi Clinical Stage 1B, 2, 3, 4 (Table 4). At these stages, lymphedema is clinically evident and not yet permanently fibrotic, sclerotic, or indurated with verrucous change.
* HIV positive
* On highly active anti-retroviral therapy
* About to initiate a course of chemotherapy
* Willingness to participate for the entire study duration, ranging from at least 14 weeks and up to 24 weeks, depending on randomization.
* Provision of written Informed Consent

Exclusion Criteria

* HIV negative
* Leg lymphedema consistent with Campisi Clinical Stage 1A or 5 (Table 4). At these stages, lymphatic dysfunction is not yet clinically evident (Stage 1A) or lymphedema has become permanently fibrotic, sclerotic, or indurated with verrucous change (Stage 5).
* History of another cancer diagnosis
* Concomitant peripheral arterial disease as documented via history or peripheral vascular physical examination
* Concomitant diagnosis of decompensated heart failure, acute phase dermatitis (at the time of the study), rheumatoid arthritis, acute phase deep vein thrombosis
* Diagnosis of medical conditions that may also lead to lower extremity lymphedema, including: congestive heart failure, filiariasis, previous vein stripping or peripheral vascular surgery
* Current use of medications known to cause edema, (i.e. calcium channel blockers, systemic corticosteroids)
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Complete Resolution of ulcers (Chronic Leg Ulcer Evaluation) | 3 years
  Proportion of completely healed ulcers at 12 weeks. The unit is number of patients with an ulcer, not number of ulcers.
Change in Lower Extremity Lymphedema Index (LELI) for KS | 3 years
  The Lower Extremity Lymphedema Index (LELI) is calculated by taking the sum of the squares of the circumference in 5 areas of a lower extremity and dividing it by the BMI. The LEL indices are significantly correlated with clinical stages and can be used as a severity scale. The LELI will compared at numerous time points throughout the study with the change in week 0 and week 14 being compared between the two arms.

SECONDARY OUTCOMES:
Time elapsed between start of wound care and complete healing of wound (Chronic Leg Ulcer Evaluation) | 3 years
  This will be assessed for the observational assessment of chronic leg ulcers
Pain and itch assessment using the Numerical Rating Scale (Chronic Leg Ulcer Evaluation) | 3 years
  Changes in the Numerical Rating Scale will be Evaluated over the period of evaluation. This marker has been previously validated in the Kenyan setting we work in.
Ability to work (Chronic Leg Ulcer Evaluation) | 3 years
  The time to improvement that facilitates work will be evaluated over the course of the observational assessment
Ability to perform household tasks (Chronic Leg Ulcer Evaluation) | 3 years
  The time to improvement that facilitates completion of household duties will be evaluated over the course of the observational assessment
Lymphedema Quality-of-Life measure (LYMQOL) for Kaposi Sarcoma | 3 years
  The Lymphedema Quality-of-Life measure (LYMQOL) has separate tools for assessing arm lymphedema and leg lymphedema. This will be compared across the two arms of the study
Change in EORTC in Kaposi Sarcoma | 3 years
  The change in the EORTC QLQ C30 (overall health quality of life in cancer patients) will be used to compare changes from Week 0 to Week 14 between immediate intervention and delayed arm. The EORTC QLQ-C30 is a questionnaire developed by the European Organization for Research and Treatment of Cancer to assess the quality of life of cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Sonak D Pastakia, PharmD,PhD, Principal Investigator — Purdue University
Locations (2):
- Kenya (2):
  - Chulaimbo District Hospital, Chulaimbo, Nyanza
  - Moi Teaching and Referral Hospital, Eldoret, Uasin Gishu County

IPD SHARING:
Plan to Share IPD: No
We don't intend to share this information unless there is a compelling, patient centered reason for sharing this information.

REFERENCES:
- [Derived] Chang AY, Karwa R, Odhiambo H, Were P, Fletcher SL, Tonui EC, Kohn MA, Lee J, Chang D, Lensing S, Namaemba DF, Busakhala N, Kiprono SK, Maurer T, Goodrich S, Pastakia SD. Compression Therapy for HIV-Associated Kaposi Sarcoma Leg Lymphedema: Results of the Kenyan Improvised Compression for Kaposi Sarcoma Randomized Controlled Trial. JCO Glob Oncol. 2022 Jan;8:e2100329. doi: 10.1200/GO.21.00329. PMID 35025687
- [Derived] Chang AY, Karwa R, Busakhala N, Fletcher SL, Tonui EC, Wasike P, Kohn MA, Asirwa FC, Kiprono SK, Maurer T, Goodrich S, Pastakia SD. Randomized controlled trial to evaluate locally sourced two-component compression bandages for HIV-associated Kaposi sarcoma leg lymphedema in western Kenya: The Kenyan Improvised Compression for Kaposi Sarcoma (KICKS) study protocol. Contemp Clin Trials Commun. 2018 Oct 21;12:116-122. doi: 10.1016/j.conctc.2018.10.003. eCollection 2018 Dec. PMID 30402565